CLINICAL TRIAL: NCT06619756
Title: Predictors of Phonological-focused Anomia Treatment
Brief Title: Anomia Treatment Predictors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Nichol Castro, Assistant Professor, State University of New York at Buffalo
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00008623
Record Dates: First submitted 2024-09-27; First posted 2024-10-01 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Anomia (Word-Finding Impairment); Aphasia
Keywords: anomia treatment; aphasia treatment
MeSH Terms: conditions — Anomia; Aphasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PMT (Experimental): Phonomotor Treatment (PMT) will be administered. This treatment improves anomia by training the sound sequences of words. This is a multimodal treatment approach that includes listening, producing, visualizing, and describing sounds and sound sequences. The participant practices the sound sequence tasks with the clinician.
  Interventions: Behavioral: Phonomotor Treatment (PMT)
- PCA (Experimental): Phonological Components Analysis (PCA) will be administered. This treatment improves anomia by identifying phonological features of words. A picture is presented. The participant provides features of the picture name: the first sound of the word, the final sound of the word, the number of syllables of the word, another word that starts with the same sound, and another words that rhymes with the word. The participant attempts to produce the word independently and by repeating after the clinician.
  Interventions: Behavioral: Phonological Components Analysis (PCA)

INTERVENTIONS:
Behavioral: Phonomotor Treatment (PMT) — Anomia treatment focuses on improving word-finding abilities. This intervention targets the phonology of words to improve word-finding.
  Arms: PMT
Behavioral: Phonological Components Analysis (PCA) — Anomia treatment focuses on improving word-finding abilities. This intervention targets the phonology of words to improve word-finding.
  Arms: PCA

SUMMARY:
The goal of this clinical trial is to identify predictors of response to phonological-focused anomia treatment in people with aphasia. The main question it aims to answer is who responds to which type of anomia treatment. Researchers will compare Phonomotor Treatment and Phonological Components Analysis to see which treatment is more beneficial, and for whom. Participants will engage in both treatments over several months.

DETAILED DESCRIPTION:
Participants will complete screening and characterization testing to determine eligibility for the study. Each treatment will be administered twice a week, for 10-15 sessions. Pre-treatment and post-treatment testing will also occur for each treatment. There will be a period of no treatment in between the first and second treatment blocks.

ELIGIBILITY:
Inclusion Criteria:

* Chronic aphasia (6+ months)
* Anomia
* Sufficient auditory comprehension to follow task instructions
* Phonologic impairment

Exclusion Criteria:

* Progressive neurological illness or disease, including dementia
* Chronic medical illness that interferes with adherence to testing schedule
* Severe, uncorrected vision or hearing impairment that interferes with task completion
* Moderate-severe apraxia of speech or dysarthria that interferes with task completion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2024-09-18 (Actual); Primary Completion 2025-10-01 (Actual); Study Completion 2025-10-01 (Actual)

PRIMARY OUTCOMES:
Naming of Trained Words | Pre-treatment and Immediately post-treatment
  Picture naming of trained words

SECONDARY OUTCOMES:
Naming of Untrained Words | Pre-treatment and Immediately post-treatment
  Picture naming of untrained words
Standardized Assessment of Phonology in Aphasia (SAPA) | Pre-treatment and Immediately post-treatment
  The SAPA assesses phonological processing abilities, including oral reading, rhyme judgments, minimal pair judgments, lexical decision, blending, and parsing.
Philadelphia Naming Test | Pre-treatment and Immediately post-treatment
  The short-form of the Philadelphia Naming Test is a picture naming test of items not seen during treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Nichol Castro, PhD, Principal Investigator — SUNY at Buffalo
Locations (1):
- UB Audiology and Speech-Language Pathology Clinic, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No
Sample size is low increasing risk of identification of individuals.